CLINICAL TRIAL: NCT03451097
Title: Evaluation of Severity of Heart Failure in Children Attending Cardiology Unit, Assiut University Children Hospital
Brief Title: Classification of Heart Failure in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, abanob wadee yousef, principal investigator, Assiut University
Other Study IDs: age based ross classification
Record Dates: First submitted 2018-02-24; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: echocardiography — cardiac ultrasound

SUMMARY:
Evaluation of Severity of Heart Failure in Children Attending Cardiology Unit, Assiut University Children Hospital

DETAILED DESCRIPTION:
Heart failure (HF) has been defined as an abnormality of cardiac structure or function leading to failure of the heart to deliver oxygen at a rate commensurate with the requirements of the metabolizing tissues, despite normal filling pressures (or only at the expense of increased filling pressures). Heart failure may result from ventricular pump dysfunction, volume overload with preserved pump function, and pressure overload with preserved pump function.Determinations of the degree of heart failure severity are essential for clinical assessment and treatment evaluation. Remarkably, no readily applied standardized method of quantifying heart failure severity exists for pediatric patients. Although standard index methods from the adult population, such as the New York Heart Association Classification, have been applied to non-infant pediatric populations, none have been validated in children. The NYHA classification measures functional capacity, not heart failure severity. The NYHA classification is inappropriate for use in pediatrics because functional capacity and responses to heart failure states differ in children compared with adults. Children have markedly different cardiac physiology, clinical presentations, and compensatory mechanisms. Moreover, the etiologies of heart failure in children are very different from those in adults. For these reasons, Ross et al.,developed a scale that is useful for grading heart failure severity in infants from birth to 6 months of age but is not applicable to older children and adolescents (Original Ross Classification).

Many have since used the "Ross Classification," including Wu et al., who confirmed an incremental rise in PNE (Plasma Norepinephrine) concentrations and progressive down-regulation of β-receptor density in children with increasing Ross class. In 1994, the Canadian Cardiovascular Society's Consensus Conference statement on the "Diagnosis and Management of Heart Failure," adopted the Ross Classification as their official scoring system for children. Ross propose an age-based Ross classification using the original variables that proved to be sensitive and specific and adding the new evidence-based data. The age ranges of 0-3 months, 4-12 months, 1-3 years, 4-8 years, and 9-18 years were chosen because the variables in the classification are generally stable during these periods but vary between them. The scoring system can be used as a continuous data set for comparison with outcomes, or it can be categorized by points.

ELIGIBILITY:
Inclusion Criteria:

* Cases admitted at Pediatric Cardiology Unit, Assiut University with Heart Failure Manifestations.

Exclusion Criteria:

* Primary liver diseases.
* Hematological diseases associated with organomegaly.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Cases admitted at Pediatric Cardiology Unit, Assiut University with Heart Failure Manifestations.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Severity of Heart Failure in Children Attending Cardiology Unit, Assiut University Children Hospital | baseline
  Evaluation of Severity of Heart Failure in Children Attending Cardiology Unit, Assiut University Children Hospital using Age based Ross classification